CLINICAL TRIAL: NCT06196515
Title: Evaluation of the Antibacterial Potential of Nano Calcium Hydroxide as an Intracanal Medication: A Randomized Clinical Trial
Brief Title: Anti-bacterial Potential of Nano Calcium Hydroxide as an Intracanal Medication
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Nada, official investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-041
Record Dates: First submitted 2023-12-10; First posted 2024-01-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Endodontic Disease; Pulp Disease, Dental
Keywords: intracanal medication
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nano calcium hydroxide in hydrogel form (Experimental): nano calcium hydroxide in hydrogel form is placed in the dry root canals after complete cleaning and shaping procedure.The intracanal medication will be distributed to fill the canals up to the orifice level.
  Interventions: Drug: nano calcium hydroxide
- Nano calcium hydroxide in paste form (Active Comparator): nano calcium hydroxide in paste form is placed in the dry root canals after complete cleaning and shaping procedure. The intracanal medication will be distributed to fill the canals up to the orifice level.
  Interventions: Drug: nano calcium hydroxide
- Conventional calcium hydroxide in paste form (Active Comparator): conventional calcium hydroxide in paste form is placed in the dry root canals after complete cleaning and shaping procedure.The intracanal medication will be distributed to fill the canals up to the orifice level.
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: Calcium hydroxide — placement of intracanal medication for the three groups will be done after cleaning and shaping of the root canals and it will be left for one week.
  Arms: Conventional calcium hydroxide in paste form
Drug: nano calcium hydroxide — placement of intracanal medication for the three groups will be done after cleaning and shaping of the root canals and it will be left for one week.
  Arms: Nano calcium hydroxide in hydrogel form; Nano calcium hydroxide in paste form

SUMMARY:
The aim of the study is to evaluate the anti-bacterial potential of Nano Calcium Hydroxide as an intracanal medication in primary endodontic treatment of permanent molars.

DETAILED DESCRIPTION:
This study is conducted to evaluate the bacterial reduction capability of hydrogel loaded with Nano Calcium Hydroxide and paste form of nano and conventional calcium hydroxide as an intracanal medication. The hydrogel will be synthesized in a new rapid in situ form that can turn from liquid into gel when reaching body temperature. The efficacy of bacterial reduction will be compared with Nano Calcium Hydroxide and conventional Calcium Hydroxide in paste form. The evaluation is to be done by quantitative microbiological assessment of samples which are gained from the root canal before and after intracanal medication placement in roots of permanent molars, having PAI score ≥ 2.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females.
* age range between 21-49.
* patients with no physical disability or psychological problems.
* patients presenting with single permanent molar with signs and/or symptoms of apical periodontitis, and having Periapican index ≥ 2.

Exclusion Criteria:

* pregnant women.
* patients with immune-compromised disease.
* patients with complicated systemic diseases.
* patients who took antibiotics within a period of 1 month.
* patients with known sensitivity to the medicaments or pharmaceuticals used in this study.
* Non-restorable teeth including root fractures, and/or advanced periodontal involvement.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
bacterial count | on the seventh day from intercanal medication placement appointment
  variation in bacterial count between 'nano calcium in hydrogel form' group compared with the other groups. The evaluation will be done by quantitative microbiological assessment test.
  Three microbiological samples will be collected from each patient. Sterile paper points will be used for collecting intracanal content and it will be sealed in Eppendorf tube until the samples reach laboratory center. Tubes will be labelled as following: S1 - S2 - S3 according to the stage of obtaining the sample.
  S1: will be obtained after access cavity and patency of canals S2: will be obtained by paper point that match the size of master apical file, after complete cleaning and shaping.
  S3: will be obtained on the seventh day from the intracanal placement appointment. paper points will be used after complete removal of the intracanal medication from the root canals.

SECONDARY OUTCOMES:
periapical healing | participants will be recalled after 6 months from the obturation for radiographic examination
  The participants will be recalled after at least 6 months, and radiographic examination of the treated tooth will be performed. Preoperative and recall radiographs of teeth will be each assigned a PAI score by 2 blinded, independent, and calibrated examiners according to Periapical index score (PAI) :
  * PAI 1: Normal periapical structure.
  * PAI 2: Bone structural changes indicating but not pathognomonic for apical periodontitis.
  * PAI 3: Bone structural changes with some mineral loss characteristic for apical periodontitis.
  * PAI 4: Well-defined apical radiolucency.
  * PAI 5: Radiolucency with radiating expansion of bone structural changes.
incidence and intensity of pain | Pain intensity will be assessed each day for three days following initial treatment
  patients will receive visual analogue scale (VAS) to help them assess pain presence and intensity each day for the following three days after intracanal placement appointment (after 24 hours, 48 hours, and 72 hours)
incidence of flare up | incidence of flare up will be recorded each day after the intracanal medication placment visit until the next visit (after seven days)
  Flare up will be presented by 'yes' for developing swelling, and 'no' for not developing swelling. it will be recorded on a chart that will be given to the patients after the initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shehab Eldin M Saber, doctoral, Study Director — British University In Egypt
Locations (1):
- british university in Egypt - dentistry collage, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No